CLINICAL TRIAL: NCT00951548
Title: Food Supplementation With the Probiotic Preparation VSL#3 as a Support to Standard Pharmaceutical Therapy in Patients With Mild to Moderate Active Ulcerative Colitis. A Double-blind, Randomized, Placebo Controlled Study
Brief Title: Food Supplementation With VSL#3 as a Support to Standard Pharmaceutical Therapy in Ulcerative Colitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VSL Pharmaceuticals (Industry)
Responsible Party: Prof. Claudio De Simone, VSL Parmaceuticals
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: VSL-UC-03
Record Dates: First submitted 2009-08-02; First posted 2009-08-04 (Estimated); Last update posted 2009-08-04 (Estimated); Status verified 2009-08

CONDITIONS: Ulcerative Colitis
Keywords: Probiotics; VSL#3; Double-blind; Placebo controlled
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- VSL#3 (Experimental): Probiotic preparation VSL#3
  Interventions: Dietary Supplement: VSL#3
- placebo (Placebo Comparator): Corn Starch
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: VSL#3 — Probiotic blend of 8 different strains of lactobacilli and bifidobacteria, dosed at 900 billion bacteria/sachet). Dosage regimen is 2 sachets b.i.d. for 8 weeks
  Arms: VSL#3
Dietary Supplement: Placebo — Corn Starch. Dosage regimen is 2 sachets b.i.d. for 8 weeks
  Arms: placebo

SUMMARY:
This is a double-blind, randomized, placebo controlled study to assess the beneficial effects of food supplementation with VSL#3 as a support to standard pharmaceutical therapy in patients affected by mild to moderate active ulcerative colitis.

DETAILED DESCRIPTION:
Title:

Food supplementation with the probiotic preparation VSL#3 as a support to standard pharmaceutical therapy in patient with mild to moderate active Ulcerative Colitis. A double-blind, randomized, placebo controlled study.

Study Design:

Double blind, randomised, parallel groups, placebo controlled, multicentre, national study.

Study Period:

February 2006 - October 2007 (recruitment: 12 months; food supplementation with VSL#3: 8 weeks).

Study Population:

The study population will comprise 144 patients with mild to moderate active ulcerative colitis on top of standard pharmaceutical therapy. 72 patients will be randomised to receive food supplementation VSL#3 and 72 to receive placebo.

Total Number of centers:

Approximately 16

Study Objectives:

To assess the beneficial effects of food supplementation with VSL#3 in patients affected by mild to moderate active ulcerative colitis in a double-blind, placebo-controlled study.

Study product:

VSL#3 consists of sachets each containing 900 billion viable lyophilised bacteria, comprising 4 strains of Lactobacillus (L. paracasei, L. plantarum, L. acidophilus and L. delbrueckii subsp. bulgaricus), 3 strains of Bifidobacterium (B. longum, B. breve and B. infantis) and 1 strain of Streptococcus thermophilus, in maltose and silicon dioxide as excipients.

The placebo is in the form of identical sachets containing only maltose and silicon dioxide.

The dose which will receive each patients is two sachets of VSL#3 or placebo to take twice a day orally (total amount of bacteria: 3.600 billion organisms per day).

Assessments:

Primary Outcome The primary outcome is the evaluation of the beneficial effects of food supplementation with VSL#3 in patients affected by UC, assessed by a decrease in the UCDAI of 50% or more, from baseline to week 8.

Secondary Outcomes:

Assessment of the beneficial effects of the food supplementation with the probiotic preparation VSL#3 on:

* activity of ulcerative colitis.
* change in subjective symptoms (rectal bleeding and stool frequency) from baseline to weeks 2, 4 and 8 of food supplementation with VSL#3.
* lack of beneficial effects, defined by need for further food supplementation or inability to stay on study till week 8.
* quality of life questionnaire (IBDQ)
* concordance between the Physician and Patient Global Assessment Scale at each time point.

Physical Status Evaluations:

Assessment of haematological laboratory tests, vital signs (blood pressure, pulse rate and respiratory rate), medical history and physical examination.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patients aged more than 18 years;
2. Diagnosis of ulcerative colitis established by previous colonoscopy, with consistent histology and clinical course;
3. Ulcerative colitis extending for more than 15 cm from the anal verge, that is involving at least the rectosigmoid. This is based on colonoscopy at any time since the onset of ulcerative colitis. Activity (not extent) must be confirmed by colonoscopy at the beginning of the study;
4. Mild to moderate active ulcerative colitis. Patients must have a minimum score of 3 and a maximum score of 8 on the 12 point UCDAI (Ulcerative Colitis Disease Activity Index - see Appendix 3) that measures stool frequency, rectal bleeding, endoscopic findings and physician's overall assessment of disease severity;
5. Symptomatic (current episode) for less than 4 weeks;
6. Minimum endoscopic score of 2 on the UCDAI at screening (mucosal appearance);
7. Use of oral 5-ASA at least 4 weeks prior to study entry, at same dose; and/or use of Azathioprine or 6-mercaptopurine at least 3 months prior to study entry, at same dose;
8. Negative pregnancy test on screening and agreeing to use valid contraception for the duration of the study;
9. Patient not requiring hospitalisation;
10. Willing an able to provide written informed consent

Exclusion Criteria:

1. Crohn's disease or pouchitis;
2. UCDAI greater than 8 (need for emergency surgery or presence of severe disease;
3. Use of oral steroids within the last 4 weeks prior to study entry;
4. Use of antibiotics within the last 2 weeks prior to study entry;
5. Change in dose of oral 5-ASA within the last 4 weeks prior to study entry and throughout the 8 week study period, or change in dose of oral 6-mercaptopurine and azathioprine drugs within the last 3 months prior to study entry and throughout the 8 week study period;
6. Use of rectal 5-ASA or steroids for one week before and throughout the 8 week study period;
7. Use of probiotic preparations either prescribed or over-the-counter within 2 weeks prior to study entry;
8. Use of NSAIDS for one week before and throughout the 8 week study period;
9. Significant hepatic, renal, endocrine, respiratory, neurological or cardiovascular disease as determined by the Investigator;
10. History of severe adverse reaction or known hypersensitivity to maltose and/or silicon dioxide;
11. Patient requiring hospitalisation;
12. Pregnant or lactating women, or women of child bearing potential not using an acceptable form of birth control (negative pregnancy test also required);
13. Use of any investigational drug and/or participation in any clinical trial within 3 months of entry to this study;
14. Inability to give a valid informed consent or to properly follow the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Actual)
Dates: Start 2006-10; Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
The primary outcome is the evaluation of the beneficial effects of food supplementation with VSL#3 in patients affected by UC, assessed by a decrease in the UCDAI of 50% or more | 8 weeks

SECONDARY OUTCOMES:
Activity of ulcerative colitis | 8 weeks
Change in subjective symptoms from baseline to weeks 2, 4 and 8 of food supplementation with VSL#3 | 8 weeks
Lack of beneficial effects, defined by need for further food supplementation | 8 weeks
Inability to stay on study | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Claudio De Simone, Prof., Study Director — VSL Pharmaceuticals
Locations (13):
- Italy (13):
  - U.O. di Medicina Interna Ospedaliera Policlinico di Bari, Bari
  - Reparto di Gastroenterologia ed Endoscopia Digestiva Azienda Ospedaliera Pugliese-Ciaccio, Catanzaro
  - U.O. Fisiopatologia Digestiva Azienda Ospedaliera Mater Domini Campus Universitario di Germaneto, Catanzaro
  - Dipartimento di Chirurgia Generale Servizio di Endoscopia Digestiva Ospedale Santa Maria Goretti, Latina
  - U.O. di Endoscopia Digestiva Presidio Ospedaliero San Salvatore, L’Aquila
  - Struttura Complessa di Medicina Interna Azienda Ospedaliera Villa Sofia - CTO Ospedale Villa Sofia, Palermo
  - U.O. di Nutrizione Clinica Ospedale Sant'Eugenio, Roma
  - P.O. Nuovo Regina Margherita Unità Operativa di Endoscopia e Gastroenterologia, Roma
  - Dipartimento di Medicina Interna U.O. di Gastroenterologia ed Endoscopia Digestiva Ospedale Cristo Re, Roma
  - Istituto di Medicina Interna CIC Columbus Policlinico Universitario Agostino Gemelli Università Cattolica del Sacro Cuore, Roma
  - Unità di Endoscopia Azienda Ospedaliera Sant'Andrea, Roma
  - Divisione di Gastroenterologia Istituto Clinico Humanitas, Rozzano (MI)
  - U.O.C. Endoscopia Digestiva IRCCS Ospedale Casa Sollievo della Sofferenza, San Giovanni Rotondo (FG)